CLINICAL TRIAL: NCT00545064
Title: A Multicenter, Open-Label Study To Evaluate The Tolerability Of Preservative Free Dorzolamide-Timolol Therapy In Patients Untreated With Open-Angle Glaucoma Or Ocular Hypertension And Dry Eye(s)
Brief Title: Dry Eye Study With Cosopt® Over 8 Weeks in Patients With Open-Angle Glaucoma or Ocular Hypertension (0507A-152)(COMPLETED)
Acronym: DISCOVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0507A-152; MK0507A-152; 2007_026
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — dorzolamide-timolol combination

INTERVENTIONS:
Drug: dorzolamide hydrochloride (+) timolol maleate — dorzolamide hydrochloride (2%)/ timolol maleate (0.5%) Preservative free twice a day (BID), for 8 weeks of treatment
  Other Names: MK0507A; Cosopt

SUMMARY:
To evaluate if preservative free cosopt is well tolerated in patients with Open angle glaucoma (OAG) or Ocular hypertension (OH) with dry eyes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with newly diagnosed and untreated for open-angle glaucoma or ocular hypertension with an Intra-ocular Pressure (IOP) of > 27 mm Hg (in at least one eye) and a baseline GSS SYMP-6 total score of 75 or less
* Patient is male or a female who is highly unlikely to conceive
* Patient has been recently diagnosed and is presently untreated for open-angle glaucoma or ocular hypertension with an IOP of at least 27 mm Hg in at least one eye (patient's worse eye)
* Patient already diagnosed with open-angle glaucoma or ocular hypertension and untreated for at least 30 days are eligible for the study if they have an IOP of 27 mm Hg or more in at least one eye

Exclusion Criteria:

* A history of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk by administering preservative free dorzolamide-timolol (preservative-free Cosopt®)
* The presence of any fundus pathology likely to change during the study or to influence IOP (background of diabetic retinopathy is permitted)
* Any contraindication to the use of preservative-free Cosopt® including:
* bronchospasm, including bronchial asthma or a history of bronchial asthma or chronic obstructive pulmonary disease, sinus bradycardia, second or third degree AV block, cardiac failure (grade III and IV), cardiogenic shock, severe renal impairment (serum creatinine > 150 umol/L or creatinine clearance < 30 ml/min)
* Patient on:
* carbonic anhydrase inhibitor, concomitant systemic or dermatological medication known to affect the IOP, e.g. clonidine, corticosteroids, oral beta-blocking agents. patient on a non-glaucoma medication that contains a preservative agent, i.e. benzalkonium chloride, benzododecinium bromide or stabilized oxychloro complex
* Patient with hypersensitivity to any component of preservative free dorzolamide-timolol (preservative-free Cosopt®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2007-05-23 (Actual); Primary Completion 2008-09-15 (Actual); Study Completion 2008-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hutnik C, Neima D, Ibrahim F, Scott R, Vaillancourt J, Haine D, Sampalis JS, Bastien N, Foucart S. Tolerability and effectiveness of preservative-free dorzolamide-timolol (preservative-free COSOPT) in patients with open-angle glaucoma or ocular hypertension. Clin Ophthalmol. 2010 Jul 21;4:581-90. doi: 10.2147/opth.s10337. PMID 20668720

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: MAY-23-2007
  Last patient out: OCT-15-2008
  Total number of sites: 28 sites in Canada. (Study performed in Canada only).
Groups:
- Preservative-free Dorzolamide-timolol (COSOPT®): subjects received preservative-free dorzolamide-timolol (COSOPT®) administered one drop in the affected eye two times daily
  The number of patients analyzed (n=176) differs from the initial tables because 2 patients withdrew consent and for whom no data were available at subsequent visits (only baseline characteristircs were available).
Period: Overall Study
Arm/Group | Preservative-free Dorzolamide-timolol (COSOPT®)
Started | 178
Visit 1 (Baseline) | 178
Visit 2 (Week 4) | 169
Visit 3 (Week 8) | 176 (8 patients didn't complete the 8-week period. 6 were retrieved and considered as Visit 3 (Week 8))
Completed | 170
Not Completed | 8
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 2
Not completed — did not complete course of treatment | 1
Not completed — cancel all appointments, no rebooking | 1
Not completed — inclement weather | 1

BASELINE CHARACTERISTICS:
Arm/Group | Preservative-free Dorzolamide-timolol (COSOPT®)
Number analyzed (Participants) | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 88

OUTCOME MEASURES:

1. Primary Outcome: Change in Glaucoma Symptom Scale (GSS)-SYMP-6 Score
Description: GSS-SYMP-6 measures 6 non-visual adverse symptoms related to glaucoma medications, with 10 5-point Likert scale questions. Score ranges between 0 and 100, lower scores indicating higher symptoms severity. Change equals post-baseline value minus baseline.
Time Frame: Baseline to week 8
Population: 176 patients qualified for inclusion in the intent to treat (ITT) analysis and completed the first visit. Observations on GSS-SYMP-6 were available for 114 and 111 patients at week 4 and 8 respectively
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Preservative-free Dorzolamide-timolol (COSOPT®) Week 4 | Preservative-free Dorzolamide-timolol (COSOPT®) Week 8
Number analyzed (Participants) | 114 | 111
Units on a Scale | 1.7 (16.8) | 3.2 (20.2)
Statistical Analysis 1: Comparison: Preservative-free Dorzolamide-timolol (COSOPT®) Week 8; The change is the post-baseline value minus the baseline value. Null Hypothesis: change in GSS-SYMP-6 score = 7; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Mean Difference (Net) = 3.2, 95% CI [-0.6 to 7.0], Standard Deviation 20.2
Statistical Analysis 2: Comparison: Preservative-free Dorzolamide-timolol (COSOPT®) Week 8; The change is the post-baseline value minus the baseline value. Null Hypothesis: change in GSS-SYMP-6 = 0; Test type: Superiority or Other; p = 0.097, t-test, 2 sided; Mean Difference (Net) = 3.2, 95% CI [-0.6 to 7.0], Standard Deviation 20.2

2. Other Pre Specified Outcome: Patient's Global Satisfaction
Description: At week 8, patients were asked to complete a single question describing how satisfied they were regarding with their medication, on a 5-level scale: very satisfied, satisfied, neither satisfied or dissatisfied, dissatisfied, very dissatisfied.
Time Frame: Week 8
Population: 178 - number of patients that signed the consent form and received at least one dose of study medication. The number of patients analyzed (n=176) differs from the initial tables because 2 patients withdrew consent and for whom no data were available at subsequent visits (only baseline characteristics were available).
Measure: Number; unit: Participants
Arm/Group | Preservative-free COSOPT® at Week 8
Number analyzed (Participants) | 170
Participants
  Very Satisfied | 79
  Satisfied | 65
  Neither Satisfied or Dissatisfied | 11
  Dissatisfied | 6
  Very Dissatisfied | 3
  Missing | 6

3. Other Pre Specified Outcome: Physician's Global Satisfaction
Description: At week 8, physicians were asked to complete a single question describing how satisfied they were regarding their patient's treatment, on a 5-level scale: very satisfied, satisfied, neither satisfied or dissatisfied, dissatisfied, very dissatisfied.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Preservative-free COSOPT® at Week 8
Number analyzed (Participants) | 170
Participants
  Very Satisfied | 130
  Satisfied | 52
  Neither Satisfied or Dissatisfied | 5
  Dissatisfied | 5
  Very Dissatisfied | 2
  Missing | 3

4. Other Pre Specified Outcome: Change in Intra-ocular Pressure (IOP) for Worse Eye From Baseline to Week 4 and From Baseline to Week 8, in Patients Receiving Preservative-free Dorzolamide-timolol
Description: IOP measurements using Goldmann applanation tonometry, performed by a masked physician two hours after patient was administered study medication. Change is computed as week 4 (or week 8) value minus baseline value.
Time Frame: Baseline to Week 4 and from Baseline to Week 8
Population: 176 patients qualified for inclusion in the intent to treat (ITT) analysis and completed the first visit. Observations on IOP were available for 164 and 166 patients at week 4 and 8 respectively
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Preservative-free Dorzolamide-timolol (COSOPT®) Week 4 | Preservative-free Dorzolamide-timolol (COSOPT®) Week 8
Number analyzed (Participants) | 164 | 166
mm Hg | -11.7 (5.1) | -11.5 (5.3)
Statistical Analysis 1: Comparison: Preservative-free Dorzolamide-timolol (COSOPT®) Week 8; The change is the post-baseline value minus the baseline value. Null Hypothesis: change in IOP = -4; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -11.5, 95% CI [-12.3 to -10.7], Standard Deviation 5.3
Statistical Analysis 2: Comparison: Preservative-free Dorzolamide-timolol (COSOPT®) Week 8; The change is the post-baseline value minus the baseline value. Null Hypothesis: change in IOP = 0; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Median Difference (Net) = -11.5, 95% CI [-12.3 to -10.7], Standard Deviation 5.3

ADVERSE EVENTS:
Description: As per protocol only Serious Adverse Events were systematically reported.
  The 0/0 indicates that Other (Not Including Serious) Adverse Events were not collected as per protocol.
Arm/Group | Preservative-free Dorzolamide-timolol (COSOPT®)
Serious Adverse Events (participants affected / at risk) | 3/178
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preservative-free Dorzolamide-timolol (COSOPT®) (N=178)
Cardiac disorders (Cardiac disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
Eye disorders (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.